CLINICAL TRIAL: NCT06898736
Title: Evaluation of Accuracy of Three-Dimensional Printing and Three-Dimensional Miniplates in Treatment of Anterior Mandibular Fractures: A Prospective Clinical Study
Brief Title: Three-Dimensional Printing and Three-Dimensional Miniplates in Treatment of Anterior Mandibular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Mazen Tharwat Abou Elkhier, Mazen Tharwat Abou Elkhier, principle investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3D printing and virtual plan
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Virtual Plan of Mandibular Fracture
Keywords: Virtual plan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- virual plan before and after mandibular fracture fixation (Experimental): virual plan before and after mandibular fracture fixation and 3D miniplate fixation
  Interventions: Device: 3d miniplate

INTERVENTIONS:
Device: 3d miniplate — 3d miniplate was used for mandibular fracture fixation

SUMMARY:
The primary objective of this study was to evaluate the accuracy of virtual reduction and the prebending of the 3D miniplates on printed models for fixation of anterior mandibular fractures. The secondary objective is to evaluate the bone healing of anterior mandibular reduction.

DETAILED DESCRIPTION:
The mandible is the largest and most prominent bone in the maxillofacial region. Facial fractures frequently involve the mandible. Rigid internal fixation combined with maxillomandibular fixation is the standard surgical procedure for treating mandibular fractures. Maxillofacial surgery currently makes extensive use of digital technology in areas like surgical navigation, titanium plate preforming technology, and 3D digital guide plate technology.

Monocortical miniplates that are easily adaptable are used in Champy's semi-rigid fixation technique, along with an "ideal osteosynthesis line" to counteract the developing masticatory forces. The location of the bone plate fixation must provide the fixation method that is most stable in relation to the line of tension at the base of the alveolar process. One plate is often used for fractures that are posterior to the foramen, and two plates are typically used for fractures anterior to the foramen.

Due to muscles working against each other, the anterior mandible fractures are subject to strong torsional forces. Some researchers have suggested using the three-dimensional (3D) miniplates as a viable option for fixation.

To ensure successful osteosynthesis with a minimally invasive approach, three-dimensional (3D) miniplate systems can be used. The system comprises two miniplates joined by interconnecting crossbars and fixed to the bone with monocortical screws. When placed in the fracture line, the 3D miniplate system ensures fracture stabilization, regardless of plate thickness and geometry. The placement of screws in a square pattern on either side of the fracture creates a solid platform that increases resistance to twisting and rotation of the longitudinal axis of the plate.

The stability of occlusion after using 3D miniplates may be due to the box-like configuration, providing rigid fixation of fractures that prevent Buccolingual splaying and gap formation at the fracture site and subsequent occlusal discrepancy; this is the advantage of 3D miniplates over 2D miniplates.

The surgeon is now able to use 3D segmentation and mirroring methods, which are highly effective in simulating the pre-traumatized anatomy at a minimal cost, using advanced open-source software programs.

The idea behind 3D printing in the medical industry is to take anatomical scans utilizing imaging methods like computed tomography (CT) and magnetic resonance imaging (MRI). The images from these methods will be saved in a common format, such as the Digital Imaging and Communications in Medicine (DICOM) format, and then with the aid of computer-aided design (CAD) software, a virtual 3D prototype with Standard Tessellation Language (STL) format will be created to enable 3D printing and the deposition of the material layer by layer to achieve the final structure.

Thus, in the present study, the goal was to assess the accuracy of virtual planning and pre-bent 3D miniplates in anterior mandibular fixation by comparing postoperative outcomes with preoperative virtual reduction and to evaluate the clinical outcomes and bone density after fixation with 3D miniplates.

ELIGIBILITY:
Inclusion Criteria:

* Recent anterior mandibular fractures (within one week).
* Adult patients of both genders (18-50 years old).
* Systematic healthy patients.
* Radiographic evidence of anterior mandibular fracture.

Exclusion Criteria:

* Medically compromised patients contraindicated for general anaesthesia and bone surgery.
* Comminuted fractures.
* Bilateral anterior mandibular fractures.
* Previously treated fractures.
* Pathological fractures and bone diseases.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Bone density was measured by Hounsfield units (HU) measured on CT images | 3 months
  The length and width of the mandible were measured using 3D CT scan with digital callipers in millimetres.
mandible dimensions | 3 months
  Mandibular length and width were measured using 3D CT scan with digital callipers in millimetres.

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - oral and maxillofacial department , faculty of dentistry, Alexandria university, Alexandria, Alexandria Governorate
  - oral and maxillofacial department, faculty of dentistry,Alexandria, Alexandria, Alexandria Governorate
  - Oral and Maxillofacial Department, Alexandria, Alexandria Governorate

IPD SHARING:
Plan to Share IPD: No
Due to [privacy/ethical/confidentiality] reasons, the research data are not publicly available.

REFERENCES:
- [Background] https://pmc.ncbi.nlm.nih.gov/articles/PMC10709695/
- [Background] Ponvel K, Panneerselvam E, Balasubramanian S, Krishna Kumar Raja VB. Evaluation of labial versus labio-inferior lines of osteosynthesis using 3D miniplate for fractures of anterior mandible: A finite element analysis with a pilot clinical trial. Chin J Traumatol. 2019 Oct;22(5):261-269. doi: 10.1016/j.cjtee.2019.08.001. Epub 2019 Aug 9. PMID 31493976
- [Background] Macdonald B, McAleer S, Kelly S, Chakraverty R, Johnston M, Pollock N. Hamstring rehabilitation in elite track and field athletes: applying the British Athletics Muscle Injury Classification in clinical practice. Br J Sports Med. 2019 Dec;53(23):1464-1473. doi: 10.1136/bjsports-2017-098971. Epub 2019 Jul 12. PMID 31300391
- [Derived] Abou Elkhier MT, Saber ME, Sweedan AO, Elashwah A. Evaluation of accuracy of three-dimensional printing and three-dimensional miniplates in treatment of anterior mandibular fractures: a prospective clinical study. BMC Oral Health. 2025 Apr 28;25(1):649. doi: 10.1186/s12903-025-05935-1. PMID 40296061